CLINICAL TRIAL: NCT04227717
Title: Assessment of a Custom-Built MRI Coil for Spine Radiotherapy Treatment Planning
Brief Title: Studying a New Piece of Equipment That Can Help Plan Radiation Therapy of the Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-476
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Thoracic Cancer; Spine Cancer; Thoracic Diseases; Spine Disease; Thoracic Neoplasms; Spine Metastases
Keywords: Thoracic lesions; Lumbar lesions; Sacral spine lesions; MRI Coil; spine radiotherapy; Memorial Sloan Kettering Cancer Center; 19-476
MeSH Terms: conditions — Spinal Cord Neoplasms; Thoracic Diseases; Spinal Diseases; Thoracic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Thoracic, lumbar and sacral spine lesions (Experimental): Participants will have thoracic, lumbar and sacral spine lesions
  Interventions: Diagnostic Test: MRI with custom MRI spine coil

INTERVENTIONS:
Diagnostic Test: MRI with custom MRI spine coil — Participants will undergo MRI with custom MRI spine coil

SUMMARY:
Participants will receive an MRI with a custom-built MRI coil for each participant. The purpose is to find out whether this custom-built MRI coil can help doctors see the different parts of the spine as well as or better than they can with standard CT myelograms.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years of age at the time of treatment
* Able to give informed consent
* Consented for spine stereotactic radiation therapy
* No contraindications for CT myelograms which include:

  * Allergy to CT contrast
  * Use of phenothiazines
  * Platelet count < 60,000 K/mcl
  * INR > 1.5
  * VEGF inhibitor use in the past 2 weeks prior to myelogram
  * NSAID use in the past 5 days prior to myelogram
  * Renal disease
  * Creatinine > 1.2 mg/dL
* No contraindications for MRI scans which include:

  * Newly placed glucose monitors
  * Tattoos (Tattoos for radiation therapy are allowed)
  * Presence of a cardiac pacemaker
  * Presence of an implanted cardioverter defibrillator
  * Breast tissue expander
  * Aneurysm clip
  * Any other implanted metallic (BB, bullet, shrapnel, IUD, metallic stent or filter, spinal cord simulator etc.) or electronic device which is considered MR unsafe
  * Severe claustrophobia or inability to lie flat for the duration of the study, etc.

Exclusion Criteria:

* Presence of surgical spine hardware at the region of interest
* Presence of cervical spine lesions
* History of claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Difference of calculated doses to the cauda equine and spinal cord based upon MRI coil vs CT myelogram used to define each structure | 6 months
  The calculated doses to the cauda equine and spinal cord will be compared and evaluated for significant difference based upon the imaging modality (MRI coil vs CT myelogram) used to define each structure, with all other target and avoidance volumes being equal in the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiya Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org